CLINICAL TRIAL: NCT02012946
Title: Levosimendan Versus Dobutamine in Cardiopatic Patients Undergoing Major Non Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, francesco pugliese, professor, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: levodobu
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Simendan; Dobutamine

ARMS (2):
- dobutamine (Active Comparator): patient receiving dobutamine
  Interventions: Drug: Dobutamine
- Levosimendan (Active Comparator): patient receiving levosimendan
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — patient receiving levosimendan
  Arms: Levosimendan
Drug: Dobutamine — patient receiving dobutamine
  Arms: dobutamine

SUMMARY:
This study wants to investigate the hemodynamic changes in cardiopatic patients undergoing major non cardiac surgery, during and after the continuous infusion of levosimendan or dobutamine.

ELIGIBILITY:
Inclusion Criteria:

* EF < 40%, no liver and renal disfynction, chronic cardiopathy

Exclusion Criteria:

* acute coronary syndrome, life expectation <30 days, hemodialysis, ventricular tachycardia/ventricular fibrillation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cardiac index | 1-3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Pugliese, Rome, Rome, Italy